CLINICAL TRIAL: NCT03522272
Title: Effectiveness of an Ultrasonic Denture Hygiene Intervention Program Among Community-dwelling Elders
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Otto Lok-Tao Lam, Clinical assistant professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UW16-266
Record Dates: First submitted 2018-04-30; First posted 2018-05-11 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-04

CONDITIONS: Denture; Removable Partial Denture; Denture Cleansers; Cetylpyridinium Chloride
Keywords: denture; removable partial denture; denture cleansers; ultrasonics; cetylpyridinium chloride; Staphylococcus aureus; Gram negative bacilli; Candida; yeast
MeSH Terms: conditions — Staphylococcal Infections; Torulopsis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ultrasonic cleaning with cetylpyridinium chloride (Experimental): Mechanical cleaning of the RPD with a soft toothbrush and liquid detergent, and ultrasonic cleaning (frequency 42kHz) (for 7 minutes 30 seconds) of the denture with 0.07% cetylpyridinium chloride mouthrinse
  Interventions: Device: Ultrasonic cleaning
- Ultrasonic cleaning with water (Active Comparator): Mechanical cleaning of the RPD with a soft toothbrush and liquid detergent, and ultrasonic cleaning (frequency 42kHz) (for 7 minutes 30 seconds) of the denture with distilled water
  Interventions: Device: Ultrasonic cleaning
- Conventional denture hygiene (Active Comparator): Mechanical cleaning of the RPD with a soft toothbrush and liquid detergent (Control group)
  Interventions: Other: Conventional denture hygiene

INTERVENTIONS:
Device: Ultrasonic cleaning — Ultrasonic cleaning (frequency 42kHz) (for 7 minutes 30 seconds) with cetylpyridinium chloride
  Arms: Ultrasonic cleaning with cetylpyridinium chloride
Device: Ultrasonic cleaning — Ultrasonic cleaning (frequency 42kHz) (for 7 minutes 30 seconds) with water
  Arms: Ultrasonic cleaning with water
Other: Conventional denture hygiene — Mechanical cleaning of denture with a soft toothbrush and liquid detergent
  Arms: Conventional denture hygiene

SUMMARY:
Objectives: The objective of this study was to assess prospectively the effectiveness of ultrasonic denture hygiene interventions in improving denture cleanliness among community-dwelling elders. Methods: A randomized clinical trial was conducted among community-dwelling elders, in which a total of 66 subjects who received upper metal framework removable partial dentures in the past five years were recruited randomly from a computerized database. They were randomly allocated into three denture hygiene intervention groups: group 1 (mechanical cleaning with a toothbrush and ultrasonic cleaning with cetylpyridinium chloride mouthrinse), group 2 (mechanical cleaning with a toothbrush and ultrasonic cleaning with distilled water) and control (mechanical cleaning with a toothbrush only). Denture cleanliness was assessed at baseline and one month review using: i) Denture Cleanliness Index (DCI) scores; ii) plaque coverage percentage; and (iii) microbiological tests. Results: There were significantly greater reductions in mean DCI scores and mean percentage of plaque coverage area in group 1 and group 2 compared to the control group for both CoCr and acrylic fitting surfaces (p<0.001). Group 1 had significant reductions in the viable counts of bacteria (CoCr and acrylic) and yeast (CoCr only) (p<0.05), while only significant reductions in bacterial viable counts (CoCr and acrylic) (p<0.05) were documented in Group 2. No significant differences were detected between groups 1 and 2 with regards to all clinical and microbiological outcomes. When comparing these parameters for CoCr and acrylic surfaces, no significant differences were observed following the intervention period. Conclusions: The ultrasonic cleaner was significantly more effective than the control in the reduction of biofilm coverage on metal framework removable partial dentures during the one month intervention period. The adjunctive use of cetylpyridinium chloride with ultrasonic cleaning did not yield improved outcomes compared to water.

ELIGIBILITY:
Inclusion Criteria:

* previously provided with cobalt chromium metal framework removable partial dentures (RPDs) within the past five years at Prince Philip Dental Hospital

Exclusion Criteria:

-

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 66 (Actual)
Dates: Start 2016-06-20 (Actual); Primary Completion 2017-06-20 (Actual); Study Completion 2017-06-20 (Actual)

PRIMARY OUTCOMES:
Denture hygiene (visual assessment) | one month
  Denture Cleanliness Index (visual assessment)

SECONDARY OUTCOMES:
Denture hygiene (planimetric assessment) | one month
  Quantitative analysis of denture cleanliness was determined by obtaining photographic images and planimetric assessment
Gram negative bacilli | one month
  Viable counts of aerobic and facultatively anaerobic bacteria
Yeasts | one month
  Viable counts of yeasts
Staphylococcus aureus | one month
  Viable counts of Staphylococcus aureus